CLINICAL TRIAL: NCT02621840
Title: A Proposed Intervention to Decrease Resident-Performed Cataract Surgery Cancellation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 14-414; 15072 (Other Grant/Funding Number: Wills Eye Hospital Innovation Grant)
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2015-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will be mandated to complete the PAT with Dr. Koka. After scheduling the surgery with the surgical coordinator, intervention patients will be required to go directly to Dr. Koka's office, to complete all necessary pre-operative steps.
  Interventions: Behavioral: Mandatory On-Site Pre-Admission Testing
- Usual Care (No Intervention): Patients in the usual care group will be treated with the standard protocol that is currently utilized in the Wills Eye Hospital Cataract and Primary Eye Care (CPEC) Service. After scheduling the surgery with the surgical coordinator, the patient will be given pre-admission testing (PAT) paperwork to be completed. The patient schedules the PAT on his or her own with the primary care physician.The patient will be given the information for Dr. Koka's cardiology office if he or she has any problem getting the PAT done.

INTERVENTIONS:
Behavioral: Mandatory On-Site Pre-Admission Testing
  Arms: Intervention

SUMMARY:
The investigators aim to investigate the impact of mandating on-site pre-admission testing on cataract cancellation rates in a randomized, prospective, intervention study. Cataract extraction is the most commonly performed ocular surgery making surgical training an integral component of ophthalmology residency. Patient cancellation of surgery results in a financial burden to the institution and a loss of essential educational experiences for the residents. An earlier study explored variables impacting cancellation rates and identified incomplete pre-admission testing as a major contributing factor to surgery cancellation.

Patients will be randomized to either 1) the intervention group where on-site pre-admission testing will be mandated or 2) the control group, where on-site pre-admission testing will be offered but not mandated. Cancellation rates will be collected prospectively and statistical analysis utilized to evaluate the significance of intervention.

DETAILED DESCRIPTION:
Cataract surgery is the most commonly performed eye surgery in the US, and it is vital for ophthalmology residents to have a high quality cataract surgery experience during their supervised training years. This allows trainees to feel comfortable performing ocular surgery and managing associated complications in a variety of clinical settings. Aspiring ophthalmologists desire a high level of surgical comfort and competence, and often times, prospective applicants to residency programs use the surgical volume and quality of training, particularly cataract surgery, as a surrogate measure for the overall quality of the residency program. This encourages residency programs to provide the most robust surgical experience possible.

Residency programs provide various levels of exposure to cataract surgery during training, from providing surgical stimulators to wet labs, where residents can practice surgical maneuvers on pig or cow eyes. These studies show that using such devices improve a resident's operative skill level, translating to greater efficiency and lower intra-operative complication rates. While practice through wet labs and surgical stimulation are clearly beneficial, there is no substitute for direct experience performing cataract surgery in the operating room. Complication rates in resident-performed cataract surgery were found to drop 50% after the resident's first 40 cases. A study evaluating the first 3000 phacoemulsification procedures of an experienced surgeon found a substantial decrease in the rate of major complications after the first 100 procedures. Another study investigating the first 1000 phacoemulsification cases performed by an experienced surgeon found an 8.4% decrease in both major and minor complications after the first 150 cases (9.3% to 0.9%).

Therefore, it is critical that ophthalmology residency programs provide a robust clinical cataract curriculum that affords residents the ability to maximize their surgical exposure and experience. Substantial exposure however, is prevented by the high rates of cancellation of cataract surgeries. This is a widespread phenomenon seen at various eye care institutions. A study of all eye surgeries cancelled at an ambulatory surgicenter in Boston found a 5.3% cancellation rate within 24 hours of the procedure, leading to a loss of at least $100,000 per year with 41% of cancellations considered preventable. Case cancellation data for 123 Veterans Administration (VA) facilities throughout 2006 showed a 9% cancellation rate for ophthalmic surgeries, with 35% of cancellations being due to "patient factors" followed by 28% due to "work up/medical condition change".

A prior study at Wills Eye Hospital found that out of the 1,083 surgeries scheduled through the Cataract and Primary Eye Care Clinic (CPEC) from 7/1/11 through 6/3/0/12, 319 (29.5%) were canceled. Of these cancellations, 72% were cancelled within 7 days of the procedure, not permitting enough time to reassign the operating room slot. Internal economic analysis at Wills has estimated lost reimbursement of these cancellations was $607,946, with $391,884 of the lost revenue from facility fees. Additionally, this is a relative loss of 230 resident surgical experiences or 28.75 surgeries missed per resident. Considered together, these findings mean that Wills Eye Hospital is not reaching its full clinical and economic potential in providing cataract surgery experience; more specifically, the institution is functioning at 86% of its capacity for cataract surgery procedures. It is apparent that the high rate of cataract surgery cancellation affects this teaching hospital both academically and economically. There is a cost to the residents who are losing valuable experience, the attending staff, and the institution as a whole.

The prior study also revealed that the most common reason for cataract surgery cancellation is patients' failure to complete pre-admission testing (PAT). While routine pre-operative testing is not supported in otherwise healthy patients undergoing elective non-cardiac surgeries, these tests are used to provide a baseline, elicit preventative measures and minimize post-operative risk. Improvement of the pre-admission testing process is modifiable and therefore presents an opportunity for intervention. Other modifiable reasons for cancellation include lack of transportation, and failure to remember not to eat the night before the procedure.

Past experience at Wills indicates that there are roughly 1100 resident cataract surgeries scheduled each year. The cancellation rate for a similar period of time determined from Assessing Cancellation Rates and Barriers to Completion of Resident Performed Cataract Surgery at Wills Eye Hospital was 29.45%, or approximately 320 cancellations per year. The investigators propose to test an intervention to address these modifiable reasons for cancellation.

Patients will be randomized to either 1) the intervention group where on-site pre-admission testing will be mandated or 2) the control group, where on-site pre-admission testing will be offered but not mandated. The intervention will be coupled with personalized patient communication appropriately timed before the scheduled procedure. Multiple studies have shown that scheduled pre-operative visitation and assessment and enhanced communication between the physician and the patient contribute to decreased cancellation of surgeries. It has been found that anesthesia-run pre-operative clinic visits significantly decrease cancellations and delays of same-day surgeries. Additionally, older patients were found to have the greatest decrease in cancellation rates after preoperative anesthesia clinic visits. At VA facilities throughout America, surgeons at low cancellation rate sites reported higher use of written preoperative instructions and pre-operative clinic visits. Cancellation rates will be collected prospectively and statistical analysis utilized to evaluate the significance of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for cataract surgery in the resident CPEC clinic at Wills Eye Hospital from the time period of 1/5/15 to 11/30/15.

Exclusion Criteria:

* All prisoners, nursing home, dialysis patients, and patients under 18 years of age will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cataract Surgery Adherence Rate | Through study completion, an average of 1 year
  The adherence rate to cataract surgery will be assessed in the usual care and intervention groups and compared.

SECONDARY OUTCOMES:
Correlation between Cataract Surgery Adherence and Demographic/Clinical Characteristics | Through study completion, an average of 1 year
  The relationship between patients' demographic/clinical characteristics and patients' adherence rates will be assessed.
Cost Analysis | Through study completion, an average of 1 year
  A cost analysis will be performed to estimate revenue losses from cancelled surgical procedures and compare costs to the previous CPEC Innovation grant, "Assessing Cancellation Rates and Barriers to Completion of Resident Performed Cataract Surgery".

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bailey, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript is under development.